CLINICAL TRIAL: NCT02369809
Title: International Postmarketing Surveillance Study of Pl-VEGF165 Safety and Efficacy in 210 Patients With Peripheral Arterial Disease
Brief Title: Non-Interventional Post Marketing Surveillance Study of Neovasculgen® in Patients With Chronic Lower Limb Ischemia
Acronym: NVG-LIGHT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Artgen Biotech (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NVG-03
Record Dates: First submitted 2015-02-17; First posted 2015-02-24 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2015-02

CONDITIONS: Lower Limb Ischemia
Keywords: Ischemia
MeSH Terms: conditions — Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neovasculgen® (Experimental): Single group prospective treatment
  Interventions: Drug: Neovasculgen®
- standard care (Active Comparator)
  Interventions: Drug: Neovasculgen®

INTERVENTIONS:
Drug: Neovasculgen® — Treatment according to routine clinical practice at the discretion of the treating physician. Patients receive two local intramuscular injections of Neovasculgen® at a course dose of 2.4 mg according to the summary of product characteristics (SmPC).
  Other Names: Neovasculgen

SUMMARY:
Aim of the study is to gain more knowledge about efficacy and safety of Neovasculgen® in daily clinical practice and obtain information about the quality of life in patients treated with Neovasculgen®.

DETAILED DESCRIPTION:
This is an open, controlled, prospective, comparative, multicentre study design. All patients received standard conservative therapy for chronic limb ischemia without cilostazol and prostaglandins and without surgical or endovascular vessel reconstruction. Surgical and endovascular vessel reconstruction was unsuitable for all of the patients

ELIGIBILITY:
Inclusion Criteria:

* Male or female person aged 40 or older
* Subject with diagnosed lower limb ischemia (Fontaine-Pokrovsky Stages IIa-III of chronic limb ischemia)
* Signed informed consent

Exclusion Criteria:

* Any disease that can, in the opinion of the treating physician, affect the outcome of the study
* Patients with addictive disorders or substance abuse
* Pregnancy or nursing
* All other exclusion criteria listed in the summary of product characteristics (SmPC)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2012-09; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change in the measurement of pain-free walking distance (PWD) on treadmill | 3 months and 6 months after the first injection of Neovasculgen®.

SECONDARY OUTCOMES:
Number of adverse drug reactions (ADRs) and unexpected adverse drug reactions (UADRs) | From the first injection of Neovasculgen® until six months after the secondary injection of Neovasculgen®
Change in the ankle-brachial index (ABI) after injection of Neovasculgen® | 3 months and 6 months after the first injection of Neovasculgen®
Change in blood flow linear velocity (BFLV) after injection of Neovasculgen® | 3 months and 6 months after the first injection of Neovasculgen®
Change in transcutaneous oxygen tension measurements (TcPO2) after injection of Neovasculgen® | 3 months and 6 months after the first injection of Neovasculgen®

CONTACTS AND LOCATIONS:
Overall Officials: Roman V Deev, MD, Study Director — +7 495 646 80 76
Locations (30):
- Russia (30):
  - "Clinical Hospital Station Barnaul Joint Stock Company" Russian Railways ", Non-governmental Health Care Institution, Barnaul, Altayskiy Kray
  - State Institution of Health Amur Region "Amur Regional Clinical Hospital", Blagoveshchensk, Amur Oblast
  - City Clinical Hospital # 21 Ufa, Ufa, Bashkortastan
  - State Budgetary Healthcare Institution "Republican Clinical Hospital Named after N.A Semashko ", Ulan-Ude, Buryatiya Republic
  - Municipal Budget Health Care Institution "City Clinical Hospital № 8". Chelyabinsk, Chelyabinsk, Chelyabinsk Oblast
  - Autonomous Healthcare Institution "Irkutsk Clinical Hospital #1 ", Irkutsk, Irkutsk Oblast
  - State Institution of Health Irkutsk "Badge of Honor" Regional Hospital, Irkutsk, Irkutsk Oblast
  - State Institution of Health of Kemerovo Region "Kemerovo Regional Hospital", Kemerovo, Kemerovo Oblast
  - Russian Academy Of Medical Sciences. Reserch Institute For Complex Problems Of Cardiovascular Diseases, Kemerovo, Kemerovskaya
  - Regional State Budget Institution of Additional Professional Education "Institute of Institute for Advanced Studies of Health Professionals" of the Ministry of Health of the Khabarovsk Region, Khabarovsk, Khabarovskiy Kray
  - State Institution of Health of the Tyumen region "Regional Clinical Hospital #1", Tyumen, Khanty-Mansiysk District
  - Regional Clinical Hospital #1 Named after Prof. S.V.Ochapovskogo of the Ministry of Health of Krasnodar Region, Krasnodar, Krasnodarskiy Kray
  - Municipal Budget Health Institution "City Clinical Hospital of Emergency Medical Care Named after N.C Karpovich ", Krasnoyarsk, Krasnoyarsk Region
  - Republican Clinical Hospital, Yoshkar-Ola, Mari El Republic
  - Federal State Institution "GBUZ MO MONIKI Named after M.F. Vladimirskogo ", Moscow, Moscow Oblast
  - State Institution of Health of Novosibirsk Region "City Clinical Hospital #1", Novosibirsk, Novosibirsk Oblast
  - Federal State Institution "Research Institute of Clinical and Experimental Lymphology", Novosibirsk, Novosibirsk Oblast
  - Budget Health Care Institution of Omsk Region "Regional Hospital", Omsk, Omsk Oblast
  - Public Health Institution "Primorsky Regional Clinical Hospital #1",, Vladivostok, Primorskiy (Maritime) Kray
  - State Educational Institution of Higher Professional Education "Rostov State Medical University", Rostov-on-Don, Rostovskaya
  - State Budgetary Healthcare Institution "Samara Regional Clinical Hospital Named after M.I. Kalinin ", Samara, Samara Oblast
  - Budgetary State Institution Samara Region Hospital # 2 Named after V.V. Banykin, Tolyatti, Samara Rigion
  - St. Petersburg Research Institute of Emergency Care named after I.I. Dzhanelidze, Saint Petersburg, Sankt-Peterburg
  - Sverdlovsk Regional Clinical Hospital #1, Yekaterinburg, Sverdlovsk Oblast
  - Public Health Autonomous Institution "Republican Clinical Hospital of the Ministry of Health of the Republic of Tatarstan", Kazan', Tatarstan Republic
  - Budgetary State Institution "Regional Hospital", Tver', Tver Oblast
  - Voronezh State Medical Academy Named After N.N Burdenko, Voronezh, Voronezh Oblast
  - State Institution of Health "Salekhard District Hospital", Salekhard, Yamal-Nenets
  - State Institution of Health Yaroslavl Region "Clinical Hospital # 10", Yaroslavl, Yaroslavl Oblast
  - State Health Care Institution "Regional Clinical Hospital", Chita, Zabaikalskii Region

REFERENCES:
- [Background] Deev R, Plaksa I, Bozo I, Isaev A. Results of an International Postmarketing Surveillance Study of pl-VEGF165 Safety and Efficacy in 210 Patients with Peripheral Arterial Disease. Am J Cardiovasc Drugs. 2017 Jun;17(3):235-242. doi: 10.1007/s40256-016-0210-3. PMID 28050885